CLINICAL TRIAL: NCT01511328
Title: Randomized Implementation of Primary Human Papillomavirus (HPV) Testing in the Organized Screening for Cervical Cancer in Stockholm
Brief Title: Randomized Implementation of Primary HPV Testing in the Organized Screening for Cervical Cancer in Stockholm
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Joakim Dillner, MD, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: SLL-KI-HPV
Record Dates: First submitted 2011-12-20; First posted 2012-01-18 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: High-grade Cervical Intraepithelial Neoplasia; Invasive Cervical Cancer
Keywords: HPV testing; Primary screening; Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HPV testing (Experimental): Women randomised to this arm get primary HPV testing
  Interventions: Other: HPV testing
- cytology (No Intervention): women included follow the standard procedure with primary cytology

INTERVENTIONS:
Other: HPV testing — Testing for Human Papilloma Virus
  Arms: HPV testing

SUMMARY:
The purpose is to evaluate whether implementation of primary human papillomavirus (HPV) screening in the screening programme for cervical cancer improves the programme in terms of better cancer protection and better cost efficiency.

DETAILED DESCRIPTION:
Primary HPV screening is a method with higher sensitivity than cytology for detection of high-grade cervical intraepithelial neoplasia, which is the precursor of cervical cancer. In particular, HPV test is a better test for revealing adenocarcinomas, since these cancers often show a normal cytology.

Cytology is less effective in older women, and screening with cytology in women over 60 has no documented effect. Today a large part of cervical cancer develop in women older than 60, to whom no screening is offered. The prevalence of HPV is around 4% in this age group. Since we know that testing negative for HPV gives a better long-term protection against cervical cancer compared to cytology, primary screening for HPV in 60-year old women would give a longer lasting protection in this high-risk group compared with today.

HPV screening is most cost effective above 35 years of age. The reason for this is that HPV is less prevalent at age 35 than in younger women and also because cervical cancer seldom develops before this age. Since the HPV test has a negative predictive value (NPV) of almost 100% this could lead to longer screening intervals, which would be improve cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

Women between the age 30 and 64 years resident in the Stockholm-Gotland region. No exclusion criteria.

Ages: 30 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 270000 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Cervical intraepithelial neoplasia 2+ (CIN2+) | first evaluation, the 1 of january 2013
  The number of women with CIN2+ detected by primary HPV testing will be compared with the number of women with CIN2+ detected by primary cytology

SECONDARY OUTCOMES:
Cost for the two different diagnostic procedures | first evaluation, 1 of January 2013
  The cost for the new procedure with HPV test in primary screening will be compared to the routine procedure with primary cytology
Invasive cervical cancer | first evaluation, after 2nd round of screening, approximately 8 years after enrollment
  The number of women with invasive cervical cancer detected in the two arms.

CONTACTS AND LOCATIONS:
Overall Officials: Joakim Dillner, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Background] Arbyn M, Ronco G, Meijer CJ, Naucler P. Trials comparing cytology with human papillomavirus screening. Lancet Oncol. 2009 Oct;10(10):935-6. doi: 10.1016/S1470-2045(09)70296-7. No abstract available. PMID 19796748
- [Background] Naucler P, Ryd W, Tornberg S, Strand A, Wadell G, Elfgren K, Radberg T, Strander B, Forslund O, Hansson BG, Hagmar B, Johansson B, Rylander E, Dillner J. Efficacy of HPV DNA testing with cytology triage and/or repeat HPV DNA testing in primary cervical cancer screening. J Natl Cancer Inst. 2009 Jan 21;101(2):88-99. doi: 10.1093/jnci/djn444. Epub 2009 Jan 13. PMID 19141778
- [Result] Lamin H, Eklund C, Elfstrom KM, Carlsten-Thor A, Hortlund M, Elfgren K, Tornberg S, Dillner J. Randomised healthcare policy evaluation of organised primary human papillomavirus screening of women aged 56-60. BMJ Open. 2017 May 30;7(5):e014788. doi: 10.1136/bmjopen-2016-014788. PMID 28566363
- [Result] Elfstrom KM, Eklund C, Lamin H, Ohman D, Hortlund M, Elfgren K, Sundstrom K, Dillner J. Organized primary human papillomavirus-based cervical screening: A randomized healthcare policy trial. PLoS Med. 2021 Aug 23;18(8):e1003748. doi: 10.1371/journal.pmed.1003748. eCollection 2021 Aug. PMID 34424907
- [Derived] Yao Q, Wang J, Elfstrom KM, Strander B, Dillner J, Sundstrom K. Evaluation of primary HPV-based cervical screening among older women: Long-term follow-up of a randomized healthcare policy trial in Sweden. PLoS Med. 2024 Dec 19;21(12):e1004505. doi: 10.1371/journal.pmed.1004505. eCollection 2024 Dec. PMID 39700313
- [Derived] Wang J, Elfstrom KM, Dillner J. Human papillomavirus-based cervical screening and long-term cervical cancer risk: a randomised health-care policy trial in Sweden. Lancet Public Health. 2024 Nov;9(11):e886-e895. doi: 10.1016/S2468-2667(24)00218-4. PMID 39486904
- [Derived] Wang J, Elfstrom KM, Lagheden C, Eklund C, Sundstrom K, Sparen P, Dillner J. Impact of cervical screening by human papillomavirus genotype: Population-based estimations. PLoS Med. 2023 Oct 27;20(10):e1004304. doi: 10.1371/journal.pmed.1004304. eCollection 2023 Oct. PMID 37889928
- [Derived] Sahlgren H, Elfstrom KM, Lamin H, Carlsten-Thor A, Eklund C, Dillner J, Elfgren K. Colposcopic and histopathologic evaluation of women with HPV persistence exiting an organized screening program. Am J Obstet Gynecol. 2020 Mar;222(3):253.e1-253.e8. doi: 10.1016/j.ajog.2019.09.039. Epub 2019 Oct 1. PMID 31585095